CLINICAL TRIAL: NCT02885051
Title: Comparative Analysis of a Behavioral Level, Skin Conductance and Heart Rate Variability in Assessing the Pain in Preterm Newborn
Brief Title: Evaluation of Pain in Preterm Newborn
Acronym: TRIPAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the end of the inclusion period, the observed correlations were much lower than expected. Thus, it did not seem relevant to prolong the inclusions.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TRIPAIN RB 16.002
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2020-10

CONDITIONS: Pain; Preterm Newborn
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preterm newborn (Experimental): Newborns hospitalized in the neonatal or Neonatal Resuscitation unit of Brest University Hospital and born before 36 weeks of gestation who will have recording of skin conductance and heart rate variability.
  Interventions: Procedure: Recording of skin conductance and heart rate variability.

INTERVENTIONS:
Procedure: Recording of skin conductance and heart rate variability. — When a procedure of care will be prescribed, installation of the electrodes of measure of the cutaneous conductance on the foot and connection of the NIPE monitor to the cardio-respiratory monitor of the child used in routine. At this stage, beginning of the video recording.

SUMMARY:
The purpose of this study is to correlate the composite PIPP-R (Premature Infant Pain Profile-Revised) scale and the parasympathetic nervous system (heart rate variability).

DETAILED DESCRIPTION:
The premature newborns hospitalized for several weeks are exposed to a significant number of nursing procedures or painful or stressful medical. Repeated pain in the neonatal period may have negative consequences in the short and / or long term. The diagnosis of pain remains difficult because based on the hetero-assessment involving the use of validated scales. The PIPP-R scale (Premature Infant Pain Profile-Revised) appears to be the most complete and best validated scale as composite (behavior items, vegetative and contextual). However, it is rarely used in routine care in France.

Alternatives to clinical scoring the pain level were described, in particular the analysis of the variability of the heart rate [VHR] by HFVI index (High Frequency Variability Index) or skin conductance. The analysis of the spectral components of high frequencies or HFVI would be an indicator of parasympathetic activity. The HFVI was compared to the EDIN scale, purely behavioral level, proposed as chronic pain marker. Skin conductance would be a stress marker reflecting variations of the sympathetic system.

These techniques are currently marketed for routine use. However, these methods have been compared and the NIPE (Newborn Infant parasympathetic Evaluation), which assesses the HFVI index, was not compared to a validated scale procedural acute pain (such as PIPP-R).

It seems important, before disseminating these methods, explore the consistency of these techniques with each other and validated scales, and their acceptability by nurses.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age less than 36 weeks
* Hospitalization in neonatology unit or intensive care unit
* Signature of major parental consent for participation of their child

Exclusion Criteria:

* Brain injury (intraventricular haemorrhage> Grade 2 or peri- ventricular leukomalacia extended)
* Administration of anticholinergic or adrenergic antagonist in the previous 48 hours
* Administration of curares
* Genetic abnormality or severe malformation

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Correlation between HFVI index and PIPP-R pain score . | 12 months plus the total duration of the patient's hospitalization
  In case of repeated measurements on the same child, only the first couple of steps will be considered for this correlation calculation.

SECONDARY OUTCOMES:
Correlation between skin conductance and pain score PIPP-R. | 12 months plus the total duration of the patient's hospitalization
  In case of repeated measurements on the same child, only the first couple of steps will be considered for this correlation calculation.
Correlation between skin conductance, HFVI and PIPP-R according to the type of painful procedure: painful or not | 12 months plus the total duration of the patient's hospitalization
  This correlation will be measured
Correlation of cutaneous conductance, HFVI and PIPP-R according to the gestational age group type | 12 months plus the total duration of the patient's hospitalization
  This correlation will be measured
Correlation of cutaneous conductance, HFVI and PIPP-R according to the sex of the child | 12 months plus the total duration of the patient's hospitalization
  This correlation will be measured
Caregiver satisfaction with each technique via the likert scale. | 12 months plus the total duration of the patient's hospitalization
  The score will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Roue, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Result] Gendras J, Lavenant P, Sicard-Cras I, Consigny M, Misery L, Anand KJS, Sizun J, Roue JM. The newborn infant parasympathetic evaluation index for acute procedural pain assessment in preterm infants. Pediatr Res. 2021 May;89(7):1840-1847. doi: 10.1038/s41390-020-01152-4. Epub 2020 Sep 22. PMID 32961546